CLINICAL TRIAL: NCT02571543
Title: Investigation of Ibuprofen in the Delay of Ovulation in NC-IVF (Natural Cycle in Vitro Fertilisation) Therapy With the Objective of Reducing Premature Ovulation and Thus Improving Effectivity (Off Label Use)
Brief Title: Can Ibuprofen Delay Ovulation in Natural Cycle-IVF?
Acronym: Ibudelay
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 015/15
Record Dates: First submitted 2015-10-07; First posted 2015-10-08 (Estimated); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Ovulation; Ovulation Inhibition; Ovulation Inhibition/Drug Effects; Pregnancy; Fertilization in Vitro/Methods
Keywords: Ibuprofen; IVF; minimal stimulation; modified natural-cycle; nonsteroidal anti-inflammatory drug (NSAID); Anti-Inflammatory Agents, Non-Steroidal/therapeutic use; Oocyte Retrieval; Ovarian Follicle/drug effects
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 2 Stage study design. Stage 1: 8 patients will be treated with the lower dose of 400mg of Ibuprofen. Should the efficacy be insufficient (3 or less patients) then the study will stop and stage 1 will recommence with 800mg.
  Stage 2: 17 patients will be treated either with the lower dose of 400mg or the higher dose of 800mg of Ibuprofen should the respective stage 1 have been successful (4 or more patients showing an effect).
  Interventions: Drug: Ibuprofen
- Control (No Intervention): The control group will consist of a no-treatment group of patients undergoing Intrauterine Insemination (IUI) or Timed Sexual intercourse (TSI), to verify the delay between LH-Peak onset and ovulation. 42h after Beta-HCG injection inducing LH-Peak, ovulation will be determined by ultrasound examination.

INTERVENTIONS:
Drug: Ibuprofen — Beginning with 400mg Ibuprofen, 5 times. Depending on the outcome of stage 1 the treatment dose will increase to 800mg, 5 times.
  Other Names: Brufen®
  Arms: Intervention

SUMMARY:
During natural cycle in vitro fertilisation, no gonadotropin stimulation is used to stimulate oocyte production. Ovulation is induced with HCG (human chorionic gonadotropin) and the follicle is retrieved 36 hours later.

In this study the patient in the intervention group will receive Ibuprofen as a study intervention beginning at the same time as the HCG injection. The treatment dose will either be 400mg every 8 to 12 hours or 800mg every 8 to 12 hours until the follicle retrieval, totalling 5 tablets. Instead of the usual time period of 36 hours, the follicular punction will occur after 42 hours. Should the oocyte still be accessible after this time period, then it is proven that Ibuprofen delays ovulation. In this case the patient will continue the regular NC-IVF treatment cycle.

The study design is a admissible two-stage design. During stage 1, 8 cycles in 8 patients will be examined. Should it be the case that after these 8 patients have completed a cycle, 4 or more show a positive treatment effect from the Ibuprofen intake, then the study will continue to stage 2 with 17 more more patients, totalling 25.

Should it be the case however, that after 8 patients, 3 or less show an effect of the Ibuprofen intake, then the study will be stopped prematurely for futility. The study intervention will be increased to 800mg of Ibuprofen and the study will recommence with 8 more patients.

A control group will consist of women undergoing intrauterine insemination (IUI) or timed sexual intercourse (TSI). 42 hours after Beta-HCG injection, an ultrasound examination will be performed in order to determine the number of remaining follicles in the ovary. This examination is to verify and control the proposed time limit of 42 hours.

DETAILED DESCRIPTION:
Background

In vitro fertilisation can be performed without the use of gonadotropin-stimulating medication, = Natural Cycle-IVF or NC-IVF for short. The effectivity of NC-IVF is limited as pro treatment cycle only one follicle develops, which can ovulate prematurely. If this is the case, a follicle aspiration is no longer possible and the next cycle must be awaited. One possibility of preventing premature ovulation is the prescription of NSAID, which is common practice in many centres, even though up until now, the effectivity has not been proven.

To test the meaningfulness of the worldwide implementation of NSAIDs in NC-IVF, a proof of concept is needed. An exactly defined study outline will explore the use Ibuprofen in a dosage of 3x400mg/24h or 3x800mg/24h. At the lower dose, Ibuprofen did not show increased side effects in randomised placebo-controlled studies.

The primary purpose of the study is therefore to determine whether or not NSAIDs in the form of Ibuprofen can successfully delay ovulation in such a way that it would be useful for everyday application in NC-IVF. Secondary purposes are to measure the effect of Ibuprofen on the Prostaglandin-E2 levels in the fluid of the extracted follicles and also whether the number of oocytes obtained in the extracted follicles differs from regular IVF-treatment.

The study design is a prospective, non-randomised, single-arm, no-treatment controlled, proof-of-concept trial. The intervention to be studied is a dose of either 400mg Brufen® or a dose of 800mg Brufen® (Drug class: Ibuprofen), taken every 8h (at night up to 12 hours) equalling a daily dose of 1200mg/24h or 2400mg/24h. The intervention will continue for 42h, totalling 5 tablets. Patients recruited will enter the study and take part for the duration of one NC-IVF treatment cycle, roughly for 2 months. Each patient can take part once, for one treatment cycle. The control group will consist of females undergoing either IUI or TSI treatment. One ultrasound examination will be performed, to measure the number of naturally occuring delayed ovulation, 42h after HCG injection. Patients recruited can take part once, for one treatment cycle.

The study population will include females between the ages of 18-42, with an indication for NC-IVF, IUI or TSI. They must wish for this treatment and fulfil all the necessary requirements, such as a regular menstruation every 26-32 days and the accessibility of both ovaries for the transvaginal follicular puncture.

The study intervention is planned with 25 completed cycles in 25 individual patients and two interim analyses which allows stopping of the trial for futility potentially after the first 8 completed cycles (two-stage design). The study control is planned with 25 treatment cycles in 25 individual patients. Blinding will not occur, as no placebo or non-historical test group will be used, thus it is an open trial.

No randomisation or stratified sampling will occur. Patients who qualify will be recruited in the NC-IVF, IUI or TSI consultations in our own Clinic.

The total study for the intervention group will span 5 consultations:

* Consult 1: Recruitment of patients, description of study and hand out of patient information informed consent documentation.
* Consult 2: Day 8-14 of the Patients' menstrual cycle. Collection of informed consent documentation and definitive enrollment in study. The patients undergo a sonographic examination of the follicle size as well as determination of E2 and LH serum levels. Following the consultation, the patients will self-inject the HCG and at the same time commence the study intervention of 400mg Brufen® every 8 hours until Consult 3.
* Consult 3: Exactly 42h after the HCG injection, the patients undergo a sonographic check of the follicle and if it remains unovulated, then it will be retrieved via vaginal access. Along with the OPU, the second study intervention in form of a 5ml venous blood sample will take place, in order to determine the serum levels of Ibuprofen.
* Consult 4: If a follicle was retrieved and successfully fertilised, 2-3 days later it will be transferred in the patients' uterus-
* Consult 5: 14-18 days after the embryo transfer, the patients will perform a pregnancy test.

Should after 8 completed cycles the dose of 400mg Brufen® not be able to show the effect of delaying ovulation in >3 of the 8 study participants, then the treatment dose will be raised to 800mg Brufen® and the study recommences.

The total study for the control group IUI will span 5 consultations:

* Consult 1: Recruitment of patients, description of study and hand out of patient information informed consent documentation.
* Consult 2: Day 8-14 of the Patients' menstrual cycle. Collection of informed consent documentation and definitive enrollment in study. The patients undergo a sonographic examination of the follicle size as well as determination of E2 and LH serum levels. Following the consultation, the patients will self-inject the HCG.
* Consult 3: Exactly 36h after the HCG injection, the patients undergo intrauterine insemination.
* Consult 4: Exactly 42h after the HCG injection, the patients undergo a sonographic check of the follicle, to see if it remains unovulated.
* Consult 5: 14-18 days after the embryo transfer, the patients will perform a pregnancy test.

The total study for the control group TSI will span 4 consultations:

* Consult 1: Recruitment of patients, description of study and hand out of patient information informed consent documentation.
* Consult 2: Day 8-14 of the Patients' menstrual cycle. Collection of informed consent documentation and definitive enrollment in study. The patients undergo a sonographic examination of the follicle size as well as determination of E2 and LH serum levels. Following the consultation, the patients will self-inject the HCG. 24-48h after HCG injection, the patients have sexual intercourse.
* Consult 3: Exactly 42h after the HCG injection, the patients undergo a sonographic check of the follicle, to see if it remains unovulated.
* Consult 4: 14-18 days after the embryo transfer, the patients will perform a pregnancy test.

Justification of the study design:

Large studies including one prospective randomised study using NSAIDs versus no medication have been performed to test the efficacy of NSAIDs. However, the study designs have been proven not to be useful to test the hypothesis that NSAIDs delay the ovulation.

Therefore the only design which will prove this hypothesis is the ovulation induction followed by a follicle aspiration so late that the follicle will definitely have been ovulated. If patients take Ibuprofen and the follicle has still not ovulated 42 hours after ovulation induction, the hypothesis will be confirmed. The time limit of 42h shall be verified by a control group, consisting of a similar patient collective as the intervention group.

Objective

* Overall Objective The purpose of this study is to evaluate whether Ibuprofen delays ovulation in such a manner that it can be used effectively in patients undergoing NC-IVF treatment and aims to describe an efficacy and safety profile for Ibuprofen in this context.
* Primary Objective The study seeks primarily to determine whether Ibuprofen can delay ovulation, in order to reduce the rate of premature ovulations in NC-IVF.
* Secondary Objectives A secondary objective is to analyse if Ibuprofen inhibits the detachment of the oocyte from the follicular wall leading to a reduced oocyte yield.

A secondary objective is to analyse the rate of delayed ovulation in the control group, after induced ovulation by HCG injection.

Methods

As a first study intervention the patient will receive 400mg of Ibuprofen every 8-12 hours until the morning of the day of the planned follicular extraction. This is the equivalent of 5 tablets beginning at the time of the HCG injection, which induces ovulation. The follicular extraction will not take place after 36 hours which is usually the case, but after 42 hours after HCG injection.

In the case of the trial being stopped for futility after the first 8 completed cycles, the treatment dose of Ibuprofen will be increased to 800mg and the study will recommence.

Should the follicle not already have ovulated then the treatment will continue as a regular IVF therapy (with the fertilisation of the oocyte and the following embryo transfer).

As a second study intervention, all patients will give a blood sample (5ml) at the time of follicle extraction in order to determine the serum concentration of Ibuprofen, thus proving that it was taken.

The control group will undergo an ultrasound examination to determine whether or not an unruptured follicle is still present in the ovary, 42h post HCG-injection.

ELIGIBILITY:
Inclusion Criteria:

* Indication for NC-IVF
* Wish for NC-IVF
* Menstruation every 26-32 days
* Accessibility of both ovaries for a follicle aspiration
* 18-42 years of age
* Written informed consent
* Indication for IUI or TSI
* Wish for IUI or TSI

Exclusion Criteria

* <18 and >42 years of age
* Gastro-intestinal diseases
* Known Ibuprofen Intolerance

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2022-08-09 (Actual)

PRIMARY OUTCOMES:
Percentage of non ovulated follicles | 42 hours after HCG injection
  The primary outcome of this study is whether Ibuprofen delays ovulation in the test subjects. It will be measured in the percentage of non-ovulated follicles exactly 42h after HCG administration with Ibuprofen.

SECONDARY OUTCOMES:
Comparison of ovulation rates between the intervention and the control groups | 42 hours after HCG injection, up to end of study duration.
  Measured using ultrasound.
Percentage of oocytes obtained from aspirated follicles | 42 hours after HCG injection
  Compared to whether this differs from regular NC-IVF without the investigational product
E2 (Estradiol) concentration in the follicular fluid | 42 hours after HCG injection
  To assess whether Ibuprofen has altered these levels
Incidence and severity of gastrointestinal and of other side effects | Throughout study duration, expected to be up to 11 months
  To assess whether Ibuprofen has caused these known side effects

CONTACTS AND LOCATIONS:
Overall Officials: Michael von Wolff, Prof. Dr., Principal Investigator — University of Bern
Locations (1):
- Department of Obstetrics and Gynecology, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Espey LL. Current status of the hypothesis that mammalian ovulation is comparable to an inflammatory reaction. Biol Reprod. 1994 Feb;50(2):233-8. doi: 10.1095/biolreprod50.2.233. PMID 8142541
- [Background] Tanaka N, Espey LL, Kawano T, Okamura H. Comparison of inhibitory actions of indomethacin and epostane on ovulation in rats. Am J Physiol. 1991 Feb;260(2 Pt 1):E170-4. doi: 10.1152/ajpendo.1991.260.2.E170. PMID 1996619
- [Background] Diao HL, Zhu H, Ma H, Tan HN, Cong J, Su RW, Yang ZM. Rat ovulation, implantation and decidualization are severely compromised by COX-2 inhibitors. Front Biosci. 2007 May 1;12:3333-42. doi: 10.2741/2316. PMID 17485303
- [Background] Gaytan M, Bellido C, Morales C, Sanchez-Criado JE, Gaytan F. Effects of selective inhibition of cyclooxygenase and lipooxygenase pathways in follicle rupture and ovulation in the rat. Reproduction. 2006 Oct;132(4):571-7. doi: 10.1530/rep.1.01236. PMID 17008468
- [Background] Gaytan M, Morales C, Bellido C, Sanchez-Criado JE, Gaytan F. Non-steroidal anti-inflammatory drugs (NSAIDs) and ovulation: lessons from morphology. Histol Histopathol. 2006 May;21(5):541-56. doi: 10.14670/HH-21.541. PMID 16493584
- [Background] Pall M, Friden BE, Brannstrom M. Induction of delayed follicular rupture in the human by the selective COX-2 inhibitor rofecoxib: a randomized double-blind study. Hum Reprod. 2001 Jul;16(7):1323-8. doi: 10.1093/humrep/16.7.1323. PMID 11425807
- [Background] Edelman AB, Jensen JT, Doom C, Hennebold JD. Impact of the prostaglandin synthase-2 inhibitor celecoxib on ovulation and luteal events in women. Contraception. 2013 Mar;87(3):352-7. doi: 10.1016/j.contraception.2012.07.004. Epub 2012 Aug 16. PMID 22902348
- [Background] Bata MS, Al-Ramahi M, Salhab AS, Gharaibeh MN, Schwartz J. Delay of ovulation by meloxicam in healthy cycling volunteers: A placebo-controlled, double-blind, crossover study. J Clin Pharmacol. 2006 Aug;46(8):925-32. doi: 10.1177/0091270006289483. PMID 16855077
- [Background] Jesam C, Salvatierra AM, Schwartz JL, Croxatto HB. Suppression of follicular rupture with meloxicam, a cyclooxygenase-2 inhibitor: potential for emergency contraception. Hum Reprod. 2010 Feb;25(2):368-73. doi: 10.1093/humrep/dep392. Epub 2009 Nov 19. PMID 19933235
- [Background] Kadoch IJ, Al-Khaduri M, Phillips SJ, Lapensee L, Couturier B, Hemmings R, Bissonnette F. Spontaneous ovulation rate before oocyte retrieval in modified natural cycle IVF with and without indomethacin. Reprod Biomed Online. 2008 Feb;16(2):245-9. doi: 10.1016/s1472-6483(10)60581-0. PMID 18284881
- [Background] Kawachiya S, Matsumoto T, Bodri D, Kato K, Takehara Y, Kato O. Short-term, low-dose, non-steroidal anti-inflammatory drug application diminishes premature ovulation in natural-cycle IVF. Reprod Biomed Online. 2012 Mar;24(3):308-13. doi: 10.1016/j.rbmo.2011.12.002. Epub 2011 Dec 15. PMID 22285246
- [Background] Rijken-Zijlstra TM, Haadsma ML, Hammer C, Burgerhof JG, Pelinck MJ, Simons AH, van Echten-Arends J, Arts JG, Land JA, Groen H, Hoek A. Effectiveness of indometacin to prevent ovulation in modified natural-cycle IVF: a randomized controlled trial. Reprod Biomed Online. 2013 Sep;27(3):297-304. doi: 10.1016/j.rbmo.2013.05.009. Epub 2013 May 22. PMID 23876971